CLINICAL TRIAL: NCT07018492
Title: A Phase 1, Open-label, Parallel-group Study to Assess the Pharmacokinetics, Safety, and Tolerability of BPN14770 in Participants With Mild, Moderate, and Severe Hepatic Impairment and Healthy Control Participants
Brief Title: Phase 1 Study of BPN14770 in Participants With Hepatic Impairment and Healthy Controls
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2414A4112
Record Dates: First submitted 2025-06-05; First posted 2025-06-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Impairment
Keywords: Mild Hepatic Impairment (HI); Moderate HI; Severe HI
MeSH Terms: interventions — BPN14770

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Mild HI (Experimental): Participants with mild hepatic impairment who have a Child Pugh classification system score of Class A will receive a single oral dose of BPN14770 capsule on Day 1.
  Interventions: Drug: BPN14770
- Group 2: Moderate HI (Experimental): Participants with moderate hepatic impairment who have a Child Pugh classification system score of Class B will receive a single oral dose of BPN14770 capsule on Day 1.
  Interventions: Drug: BPN14770
- Group 3: Severe HI (Experimental): Participants with severe hepatic impairment who have a Child Pugh classification system score of Class C will receive a single oral dose of BPN14770 capsule on Day 1.
  Interventions: Drug: BPN14770
- Group 4: Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single oral dose of BPN14770 capsule on Day 1.
  Interventions: Drug: BPN14770

INTERVENTIONS:
Drug: BPN14770 — Administered as specified in the treatment arm.

SUMMARY:
The primary purpose of this study is to assess the pharmacokinetics (PK) of BPN14770 after a single oral administration of BPN14770 in participants with mild, moderate, and severe liver impairment compared with control participants with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

* Considered to be healthy (for healthy participants) or medically stable (for participants with hepatic impairment), as determined by medical evaluation.
* Body weight ≥ 50 kilograms (kg) and body mass index (BMI) within the range ≥ 18.5 to < 40.0 kilograms per square meter (kg/m^2).
* A diagnosis of clinically stable hepatic disease for at least 1 month prior to the screening visit, confirmed by medical history or previous confirmation of hepatic cirrhosis by liver biopsy or medical imaging technique.
* Mild, moderate, and severe hepatic impairment based on the Child-Pugh classification score at the screening visit and Day ˗1 to determine eligibility:

  * Mild (Class A) hepatic impairment (Child-Pugh classification score 5 to 6)
  * Moderate (Class B) hepatic impairment (Child-Pugh classification score 7 to 9)
  * Severe (Class C) hepatic impairment (Child-Pugh classification score 10 to 15)
* Healthy Participants matched to each participant with moderate hepatic impairment with respect to sex, age (± 10 years), and BMI (± 10%)

Key Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data, in the judgment of the investigator.
* Blood loss or blood donation that exceeds 500 milliliters (mL) within 56 days prior to or at the screening visit or donation of any amount of blood from the screening visit until admission to the clinical research unit (CRU).
* Healthy participants:

  * Clinical laboratory values outside the reference range during the screening period or on Day ˗1 and considered clinically significant by the investigator
  * Alanine aminotransferase or aspartate aminotransferase > 1.5 * the upper limit of normal (ULN) or bilirubin ≥ 1.0 * the ULN.
* Participants with hepatic impairment:

  * Participant with clinically significant laboratory values in the opinion of the investigator or outside the acceptable ranges or limits during the screening period.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Time Curve Extrapolated from Time 0 to Infinity (AUCinf) of BPN14770 | Predose up to 240 hours postdose
Maximum Observed Plasma Concentration (Cmax) of BPN14770 | Predose up to 240 hours postdose
Time Maximum Observed Plasma Concentration (Tmax) of BPN14770 | Predose up to 240 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 15 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Shionogi Inc.
Locations (3):
- United States (3):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No